CLINICAL TRIAL: NCT05351931
Title: A Randomized Phase 2 Double-blind Placebo-controlled Trial Investigating the Effect of Salovum™ and SPC-flakes on Radiochemotherapy Induced Toxicity in Curative Treatment of Anal Carcinoma
Brief Title: Role of Antisecretory Factor in Curative Radiochemotherapy for Anal Carcinoma
Acronym: SALFLAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uppsala University Hospital (Other)
Collaborators: Lantmännen AB (Unknown); Sjöbergstiftelsen (Unknown); Onkologiska klinikens forskningsfond (Unknown); Swedish Cancer Society (Other)
Responsible Party: Principal Investigator, Peter Nygren, Professor, consultant in oncology, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASF 3
Record Dates: First submitted 2022-04-14; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Anal Cancer
Keywords: Radiochemotherapy; Adverse event; Antisecretory factor
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized parallel two groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo similar to active study products
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPC-flakes with or without Salovum (Active Comparator): SPC-flakes flat dose of 75 g/d divided in 2 - 4 doses started 5 days prior to start of RCT and continued during the RCT. Salovum egg powder 4 g/sachet. Four sachets, ie 16 g q 8 h for 5 days prior to start of RCT. The appropriate amount of Salovum is mixed with 100 - 200 ml of suitable liquid, eg fruit juice, and ingested orally.
  Interventions: Dietary Supplement: Salovum and SPC-flakes or corresponding placebo
- SPC-flakes placebo with or without Salovum placebo (Placebo Comparator): SPC-placebo flat dose of 75 g/d divided in 2 - 4 doses started 5 days prior to start of RCT and continued during the RCT. Salovum placebo egg powder 4 g/sachet. Four sachets, ie 16 g q 8 h for 5 days prior to start of RCT. The appropriate amount of Salovum placebo is mixed with 100 - 200 ml of suitable liquid, eg fruit juice, and ingested orally.
  Interventions: Dietary Supplement: Salovum and SPC-flakes or corresponding placebo

INTERVENTIONS:
Dietary Supplement: Salovum and SPC-flakes or corresponding placebo — Salovum and SPC-flakes are foods approved for specific medical purposes.

SUMMARY:
Curative radiochemotherapy (RCT) for anal carcinoma (AC) is associated with considerable acute and long-term toxicity. The acute toxicity derives from the combined effects of radiation and chemotherapy and is dominated by localized skin mucositis, diarrhoea and pain from radiation and nausea, fatigue, anemia/leukopenia, diarrhoea and general skin dryness from chemotherapy. Cholera induced diarrhoea, as well as other forms of diarrhoea-inducing agents, has been shown to elicit a stimulated, endogenous production of a protein, named "antisecretory factor" (ASF). This protein has been chemically characterized in detail. ASF acts by modulating secretion of water and ions but also counteracts inflammatory processes. With this background the present study will investigate if induction of endogenous ASF by intake of SPC-flakes might be beneficial in AC patients to prevent RCT induced adverse events (AEs) and if administration of ASF from Salovum provides additional benefit (explorative).

DETAILED DESCRIPTION:
Curative RCT for AC is associated with considerable acute and long-term toxicity.

The acute toxicity derives from the combined effects of radiation and chemotherapy and is dominated by localized skin mucositis, diarrhoea and pain from radiation and nausea, fatigue, anemia/leukopenia, diarrhoea and general skin dryness from chemotherapy. These adverse effects are treated symptomatically with mostly modest effect and sometimes leads to the need for in-patient care and temporary stop of the RCT. Long-term toxicity is caused by radiation fibrosis and is dominated by impaired anal sphincter function leading to faeces incontinence, pelvic pain and reduced sexual function. Thus, new ways to efficiently counteract the RCT induced adverse effects are urgently needed.

Cholera induced diarrhoea, as well as other forms of diarrhoea-inducing agents, has been shown to elicit a stimulated, endogenous production of a protein, named "antisecretory factor" (ASF). This protein has been chemically characterized in detail. ASF acts by modulating secretion of water and ions but also counteracts inflammatory processes . ASF is also produced by hens fed on a diet of fermented grains or a specific diet of sugars and amino acids, leading to an accumulation of the ASF protein in the egg yolk. Spray dried yolk in the form of a powder is commercialized as Salovum registered by the EU authorities as "Food for specific medical purposes", i e is not adrug from a regulatory perspective.

Salovum rapidly increase the plasma (P-) ASF-concentration. Another way to increase ASF and, thus, to achieve benefit, is to induce its production/conversion by ingestion of oat flakes, specially processed (similar to malting) to contain the proper mix of sugars and amino acids. Such flakes are also commercially available (named SPC flakes) as "Food for specific medical purposes" and has been recommended or considered for a number of secretory pathological conditions, e g for treatment of Mb Meniére.

With this background the present study will investigate if induction of endogenous ASF by intake of SPC-flakes might be beneficial in AC patients to prevent RCT induced adverse events (AEs) and if administration of ASF from Salovum provides additional benefit (explorative).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histologically confirmed diagnosis of AC irrespective of tumour p16-status.
3. Planned for curative RCT according to national care programme schedule B
4. WHO performance status of 0 or 1.
5. For patients planned for schedule C, they must be unsuitable for or not consenting to participation in the SWANCA trial.
6. Able to understand study information and questionnaires and provide signed informed consent.

Exclusion Criteria:

1. Patients with stoma.
2. Contraindications to the investigational product, e g known or suspected hypersensitivity to the investigational products or expected inability to their use in accordance with the protocol.
3. Contraindications to curative RCT in accordance with AC national care programme.
4. Lack of suitability for participation in the study, e g expected difficulties to follow the protocol procedures, as judged by the investigator.
5. Prior exposure to Salovum or SPC-flakes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of diarrhoea, fecal urgency, anal skin toxicity/mucositis and anal pain CTCAEv5.0 ≥ grade 2 during and up to 6 months after RCT. Anal skin toxicity/mucositis is to be verified by photos. | Through study completion, approximately 6 months
  Treatment related toxicity

SECONDARY OUTCOMES:
Incidence and severity of other AEs according to CTCAEv5.0 during and up to 6 months after RCT. | Through study completion, approximately 6 months
  Other treatment related toxicity
Change from baseline in patient reported hQoL and abdominal symptoms assessed by EORTC QLQ- 30 and the ANL27 subscale questionnaires as well as the Bristol Stool Form Scale. | Through study completion, approximately 6 months
  PROMS
Increase in plasma (P)-ASF concentration from baseline to the day of start of RCT and to the end of treatment. | Days -1, 6 and 42
  Pharmacodynamic outcome and compliance check
Relationships between P-ASF concentration, biomarkers reflecting inflammation and adverse events. | Through study completion, approximately 6 months
  Biomarker assessments
Differences in primary and secondary endpoints between Salovum and placebo subgroups. | Through study completion, approximately 6 months
  Assessment of added value of Salovum
Tumour response rate according to RECIST v1.1 and clinical examination at 2, 3 (radiology) and 6 months after stop of RCT. | Through study completion, approximately 6 months
  Assessment of benefit, if any, from study products on clinical outcome
Disease free and overall survival at 3 and 6 months after stop of RCT. | At 3 and 6 months after stop of treatment
  Assessment of benefit, if any, from study products on clinical outcome

OTHER OUTCOMES:
Incidence of AEs CTCAEv5.0 grade ≥ 2 considered probably related to investigational products/placebo. | Through study completion, approximately 6 months
  Adverse effects from study products

IPD SHARING:
Plan to Share IPD: No
To be considered

REFERENCES:
- [Background] Cinausero M, Aprile G, Ermacora P, Basile D, Vitale MG, Fanotto V, Parisi G, Calvetti L, Sonis ST. New Frontiers in the Pathobiology and Treatment of Cancer Regimen-Related Mucosal Injury. Front Pharmacol. 2017 Jun 8;8:354. doi: 10.3389/fphar.2017.00354. eCollection 2017. PMID 28642709
- [Background] Ulgheri C, Paganini B, Rossi F. Antisecretory factor as a potential health-promoting molecule in man and animals. Nutr Res Rev. 2010 Dec;23(2):300-13. doi: 10.1017/S0954422410000193. Epub 2010 Aug 5. PMID 20684797
- [Background] Johansson E, Jennische E, Lange S, Lonnroth I. Antisecretory factor suppresses intestinal inflammation and hypersecretion. Gut. 1997 Nov;41(5):642-5. doi: 10.1136/gut.41.5.642. PMID 9414971
- [Background] Lonnroth I, Lange S. Purification and characterization of the antisecretory factor: a protein in the central nervous system and in the gut which inhibits intestinal hypersecretion induced by cholera toxin. Biochim Biophys Acta. 1986 Aug 6;883(1):138-44. doi: 10.1016/0304-4165(86)90144-3. PMID 3524692
- [Background] Laurenius A, Wangberg B, Lange S, Jennische E, Lundgren BK, Bosaeus I. Antisecretory factor counteracts secretory diarrhoea of endocrine origin. Clin Nutr. 2003 Dec;22(6):549-52. doi: 10.1016/s0261-5614(03)00057-8. PMID 14613757
- [Background] Eriksson A, Shafazand M, Jennische E, Lange S. Effect of antisecretory factor in ulcerative colitis on histological and laborative outcome: a short period clinical trial. Scand J Gastroenterol. 2003 Oct;38(10):1045-9. doi: 10.1080/00365520310005064. PMID 14621278